CLINICAL TRIAL: NCT01044082
Title: Impact of Controlled Cord Traction During the Third Stage of Labour on the Incidence of Post Partum Haemorrhage
Brief Title: Prevention of Post-partum Haemorrhage
Acronym: TRACOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P081206; AOM09161 (Other Grant/Funding Number: AOM09161)
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-03

CONDITIONS: Postpartum Haemorrhage; Immediate Postpartum Hemorrhage
Keywords: Postpartum haemorrhage; Third stage of labour; Controlled cord traction; Randomized controlled trial; Prevention
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- controlled cord traction (Experimental): Controlled cord traction will be applied as soon as a firm uterine contraction is obtained, and until placental delivery occurs.
  Interventions: Procedure: controlled cord traction
- clinical signs of placental separation (Active Comparator): Clinical signs of placental separation will be awaited for, and then placental expulsion may be helped through maternal pushing and/or hypogastric pressure
  Interventions: Procedure: Clinical signs of placental separation

INTERVENTIONS:
Procedure: controlled cord traction — In the intervention group, controlled cord traction will be applied as soon as a firm uterine contraction is obtained, and until placental delivery occurs
  Arms: controlled cord traction
Procedure: Clinical signs of placental separation — Clinical signs of placental separation will be awaited for, and then placental expulsion may be helped through maternal pushing and/or hypogastric pressure
  Arms: clinical signs of placental separation

SUMMARY:
The primary purpose of the trial is to evaluate whether the management of placental delivery with controlled cord traction (CCT) reduces the incidence of postpartum haemorrhage, compared with management waiting for clinical signs of spontaneous placental separation, in women with vaginal delivery receiving prophylactic oxytocin for the management of the third stage of labour.

The hypothesis is that CCT, by reducing the length of the third stage of labour, facilitates early postpartum uterine contraction and local haemostasis and decreases post partum blood loss.

DETAILED DESCRIPTION:
In this randomized controlled trial, conducted in 6 maternity units, information will be provided to eligible women during a prenatal visit in late pregnancy. Once in labour ward, during labour and before delivery, and if eligible and willing to participate, the woman will be randomly allocated to the intervention or reference group.

In all women, immediately after the birth of the baby, 5 IU prophylactic oxytocin will be intravenously administered, the umbilical cord will be early clamped and cut, and a collector bag placed under the woman's buttocks.

In the intervention group, controlled cord traction will be applied as soon as a firm uterine contraction is obtained, and until placental delivery occurs.

In the reference group, clinical signs of placental separation will be awaited for, and then placental expulsion may be helped through maternal pushing and/or hypogastric pressure.

All other aspects of the management of the third stage will be standardized and common to all women.

On day 2 postpartum, a venous blood sample will be collected to measure plasma haemoglobin and haematocrit. On the same day, a questionnaire will be filled in by the woman to assess her satisfaction.

ELIGIBILITY:
Inclusion criteria :

* Age ≥ 18
* Expected vaginal delivery
* Gestational age ≥ 35 weeks
* Singleton pregnancy

Exclusion criteria :

* Age <18
* Planned caesarean delivery
* Severe hemorrhagic disease
* Multiple Pregnancy
* Placenta praevia
* Intra uterine fetal death
* No health insurance coverage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4382 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Incidence of postpartum haemorrhage, defined as a measured postpartum blood loss greater than 500 mL | immediately to two hours after delivery

SECONDARY OUTCOMES:
Severe postpartum haemorrhage, defined as a measured postpartum blood loss greater than 1000mL | immediately to two hours after delivery
Measured postpartum blood loss at 30 minutes after delivery | at 30 minutes after delivery
Total measured postpartum blood loss | Time after delivery
Curative postpartum uterotonic treatment | Time after delivery
Postpartum transfusion | Time after delivery
Postpartum embolization or surgery for haemorrhage | Time after delivery
Peripartum haemoglobin delta | Time after delivery
Peripartum haematocrit delta | Time after delivery
Duration of third stage of labour | time before delivery
Deliveries with manual removal of placenta | 30 minutes
Potential adverse events: uterine inversion, cord rupture, pain during third stage of labour | Time after delivery
Woman's satisfaction | two days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Deneux, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Maternité de Port-Royal, Paris, France

REFERENCES:
- [Derived] Deneux-Tharaux C, Sentilhes L, Maillard F, Closset E, Vardon D, Lepercq J, Goffinet F. Effect of routine controlled cord traction as part of the active management of the third stage of labour on postpartum haemorrhage: multicentre randomised controlled trial (TRACOR). BMJ. 2013 Mar 28;346:f1541. doi: 10.1136/bmj.f1541. PMID 23538918